CLINICAL TRIAL: NCT03180333
Title: The Tolerability and Pharmacokinetics Clinical Trial of Metacavir Enteric-coated Capsules in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangzhou Yipinhong Pharmaceutical CO.,LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PNA-20120309-V1
Record Dates: First submitted 2017-05-31; First posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- PNA 1 (Experimental): Multiple dosing tolerance test:Metacavir Enteric-coated Capsules 160mg/320mg,once a day,continuous administration for 7 days;
  Interventions: Drug: PNA
- PNA placebo (Placebo Comparator): Multiple dosing tolerance test:Metacavir Enteric-coated Capsules placebo 160mg/320mg,once a day,continuous administration for 7 days
  Interventions: Drug: PNA placebo
- PNA 2 (Experimental): Single dosing pharmacokinetic test:Metacavir Enteric-coated Capsules 80mg/160mg/320mg,single-dose;
  Interventions: Drug: PNA
- PNA 3 (Experimental): Multiple dosing pharmacokinetic test:Metacavir Enteric-coated Capsules 160mg/320mg,once a day,continuous administration for 6 days;
  Interventions: Drug: PNA
- PNA 4 (Experimental): The effect of diet:Metacavir Enteric-coated Capsules 160mg,before and after meal.
  Interventions: Drug: PNA

INTERVENTIONS:
Drug: PNA
  Other Names: Metacavir Enteric-coated Capsules
  Arms: PNA 1; PNA 2; PNA 3; PNA 4
Drug: PNA placebo
  Other Names: Metacavir Enteric-coated Capsules placebo
  Arms: PNA placebo

SUMMARY:
Conduct in Chinese healthy adult subjects:1.To observe the safety and tolerability of multiple-dose oral administration of different doses of PNA;2.By measuring the changing drug concentration in the plasma and urine after a single oral administration of different doses of PNA on the condition of fasting, the pharmacokinetic parameters of the single dose are estimated;3.By measuring the changing drug concentration in the plasma of PNA after a multiple-dose oral administration on the condition of fasting, the pharmacokinetic parameters of multiple-dose are estimated, and a basis for dosage regimens of the clinical research phase Ⅱ is provided;4.To study the effects of diet on the pharmacokinetic parameters via the changes of concentration of PNA in plasma after high-fat and high-calorie food.

DETAILED DESCRIPTION:
The study is divided into three parts:

1. The tolerance test of randomized，double-blind, placebo-controlled multiple-dose oral administrations.2 dosage groups are set up.Each group contains 8 subjects,evenly composed of men and women.The beginning dosage of the study is 160mg/L.Subjects who have successfully completed tests of the beginning dosage group and passed the safety assessment will enter the test of next dosage group(320mg/L) according to the same method.
2. Pharmacokinetic tests(single/multiple dose) .(1)Single dosing pharmacokinetic tests.36 eligible healthy subjects are selected. Each group has 12 people, evenly composed of men and women. After taking 80mg/160mg/320mg of PNA orally in fasting state, blood and urine samples are taken to be tested and analyzed, in order to study the pharmacokinetic characteristics of single-dose administrations.(2)Multiple dosing pharmacokinetic tests.In the single-dose administration trial, respectively choose 10 subjects (evenly composed of men and women) in middle and high-dose group (160mg qd、320mg qd).After the single-dose administration,inspecte the pharmacokinetic characteristics with 6-day continuous administration. Blood samples are taken to test the trough drug concentration of pre-dose in the morning of the 3rd, 4th, 5th day after administration, and the 6th morning before and after the administration, to study the steady state concentration and the fluctuation coefficient of the trough to peak drug concentration after multiple-dose, and to find out whether there exists the effect of drug storage and / or induction of drug enzyme.
3. The effect of diet.Choose 12 qualified healthy subjects (normally evenly composed of men and women), a randomized two-way cross-over design is used, respectively orally take 160 mg of PNA before and after meal, and to study the effect of diet on pharmacokinetic via blood collection.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers aged 18 to 45 years old ;
2. Body mass index (BMI) above/equal 19 and below 24 kg/m2;
3. Child bearing potential, has a negative serum pregnancy test at screening period, and agrees to use contraceptions consistently and correctly in 14 days after dosing;
4. Subjects with no cardiovascular, liver, kidney, digestive tract, nervous and mental and other acute or chronic diseases that may affect the safety and pharmacokinetic of drug;
5. Signed informed consent voluntarily.

Exclusion Criteria:

1. Subjects not meet the inclusion criteria;
2. Abnormal clinically significant laboratory results;
3. Abnormal clinically significant electrocardiogram (ECG);
4. A positive hepatitis B surface antigen, hepatitis C or HIV test result;
5. History of hypersensitivity or allergy to any of the study drugs or to drugs of similar chemical classes;
6. Addicted to smoking and drinking;
7. Drink in 36 hours before post-dosing of study drug;
8. Ingest any foods or beverages which may affect pharmacokinetics;
9. Drug abuse,a history of poisoning;
10. Subjects who had received other medications within 2 weeks prior to the first administration of Investigational Product，and the original and main metabolites were not completely eliminated ;
11. Subjects who participated in any other clinical trials within 3 months prior to the first administration of Investigational Product;
12. Subjects who had suffered from hemorrhage or blood donation over 200ml will be excluded;
13. Subjects over exercised accompanied with fatigue and muscle aches within 1 week period to the first administration of Investigational Product;
14. Children,women who are pregnant,lactating,with childbearing potential and who are using acyeterions;
15. Subjects in the opinion of the investigator, could not participate in this study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
TEAEs | day 1 to day 14
  Frequency of treatment-emergent adverse events

SECONDARY OUTCOMES:
AUC | day 1 to day 7
  Area under the plasma concentration versus time curve of PNA
Cmax | day 1 to day 7
  Maximum Plasma Concentration of PNA
T1/2 | day 1 to day 7
  The time required while plasma concentration is reduced by half of PNA

CONTACTS AND LOCATIONS:
Overall Officials: Hongwei Fan, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University; Ruifang Wang, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No